CLINICAL TRIAL: NCT00109330
Title: A Phase III, Observer-blinded Randomised, Multi-centre Clinical Study of the Safety, Immunogenicity and Consistency of Three Manufacturing Lots of GSK Biologicals' Candidate Tdap Vaccine as Compared to a US-licensed Td Vaccine When Given as a Booster Dose to Healthy Adolescents (10-18 Years of Age)
Brief Title: A Combined Tdap Vaccine Used As A Booster Compared To Licensed Td Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 776423/001
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Diphtheria; Tetanus; Acellular Pertussis
Keywords: Prevention of Diphtheria, Tetanus, Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid

INTERVENTIONS:
Biological: Combined diphtheria, tetanus, acellular pertussis vaccine

SUMMARY:
This study will evaluate the safety and immune response to GlaxoSmithKline Tdap vaccine compared to licensed Td vaccine when used as a booster in healthy adolescents (10-18 years of age).

DETAILED DESCRIPTION:
A combined Tdap (Tetanus, Diphteria, Acellular Pertussis) Vaccine Used as a Booster compared to Licensed Td (Tetanus and Diphteria) vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents with history of completed routine vaccination against diphtheria, tetanus, and pertussis (DTP).

Exclusion Criteria:

* Use of any other investigational drug or vaccine 30 days preceding study vaccination.
* Chronic administration of immunosuppressants.
* Administration of pre-school DTP vaccine within previous 5 years.
* Administration of Td booster within previous 10 years.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4116 (Actual)
Dates: Start 2002-11; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (42):
- United States (42):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Rolling Hills Est, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Yorba Linda, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Middletown, Connecticut
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, New Bedford, Maine
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Whitehouse Station, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Lumberton, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, University Heights, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 776423/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 776423/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 776423/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 776423/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 776423/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 776423/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register